CLINICAL TRIAL: NCT02033954
Title: PrOspective, MultiCenter Study for the Evaluation of PerformanCe of the ArtVentive Medical Group Peripheral EndoLuminal OcclUsion SystemTM for the Peripheral Embolization Treatment to Rapidly OccluDe Venous or Arterial BleEding - OCCLUDE II
Brief Title: Evaluation of Peripheral EOS for the Peripheral Embolization Treatment to Rapidly OccluDe Venous or Arterial BleEding
Acronym: OCCLUDE-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ArtVentive Medical Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TD 0088 / 04
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Hemorrhage; Bleeding
Keywords: Embolization; Hemorrhage; TIPS; GI Bleeding; AV Fistula; AV Malformation; Traumatic Vascular Injury
MeSH Terms: conditions — Hemorrhage; Gastrointestinal Hemorrhage; Arteriovenous Fistula; Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To collect confirmatory data in support of the safety and performance of the ArtVentive Medical Group Endoluminal Occlusion System.

DETAILED DESCRIPTION:
Prospective, non-randomized, multi-center confirmatory observational study for the treatment of subjects with the need for vascular occlusion for the following conditions:

1. Stopping blood loss from a damaged blood vessel from a traumatic vascular injury
2. Hemorrhage caused by a neoplasia
3. Neoplastic process (tumor)
4. Gastrointestinal bleeding
5. Closing an abnormal blood vessel supplying a vascular anomaly such as arteriovenous malformations or an arteriovenous fistula
6. Interrupting blood supply to an organ or part of an organ for permanent devascularization
7. Devascularization of tissues involved by a neoplastic process either pre-operatively or as a palliative measure
8. Transjugular Intrahepatic Portosystemic Shunt (TIPS)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥18 to ≤75 years.
2. Subject with target vessels of 3.0 mm to 12 mm in diameter.
3. Subject is able and willing to comply with all study requirements, including the required study follow-up visits.
4. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the consent form. In the event of emergency procedure and subject and/or legal representative is unable to provide consent prior to study enrollment, consent will be obtained at earliest possible time following procedure for consent to continue to participate in the study.

Exclusion Criteria:

1. Subject has a known allergy to iodinated contrast for which they cannot be adequately premedicated.
2. Subjects in whom venography or arteriography is contraindicated.
3. Subjects with known hypersensitivity or contraindication to nickel or nitinol.
4. Subject is pregnant or breastfeeding.
5. Any clinical evidence that the investigator feels would place the subject at increased risk with the deployment of the device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects requiring permanent occlusion of the peripheral vessels for the following conditions:
  1. Stopping blood loss from a damaged blood vessel from a traumatic vascular injury
  2. Hemorrhage caused by a neoplasia
  3. Neoplastic process (tumor)
  4. Gastrointestinal bleeding
  5. Closing an abnormal blood vessel supplying a vascular anomaly such as arteriovenous malformations or an arteriovenous fistula
  6. Interrupting blood supply to an organ or part of an organ for permanent devascularization
  7. Devascularization of tissues involved by a neoplastic process either pre-operatively or as a palliative measure.
  8. Transjugular Intrahepatic Portosystemic Shunt (TIPS)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Safety | Acute & 30 days
  Composite of new-onset major device-related adverse event(s) including device embolization beyond targeted treatment area (not therapeutic indication of embolization), need for emergency surgical intervention of the target vessel, or distal embolization (non-device embolization, e.g., particulate matter / plague distal to the device) at 30 days.

SECONDARY OUTCOMES:
Occlusion | 30 days
  Sustained occlusion at 30 days follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Mahnken, Prof Dr, Principal Investigator — Universitätsklinikum Giessen und Marburg (UKGM) Klinik für diagnostische und
Locations (7):
- Austria (2):
  - Klinikum Klagenfurt am Worthersee, Klagenfurt
  - Krankenhaus der Barmherzigen Schwestern Linz Betriebsgesellschaft m.b.H., Linz
- UZ Leuven, Leuven, Belgium
- Germany (4):
  - Universitatsklinikum Carl Gustav Carus Institut, Dresden
  - Universität Leipzig - Department für Bildgebung und Strahlenmedizin, Leipzig
  - Universitätsklinikum Giessen und Marburg (UKGM) Klinik für diagnostische und, Marburg
  - LMU Klinikum der Universität München, Campus Innenstadt, Interventionelle Radiologie, Munich

REFERENCES:
- [Background] Venbrux AC, Rudakov L, Plass A, Emmert MY, Ebner A. A new occlusion device: application of the ArtVentive endoluminal occlusion system (EOS)--first in human clinical trial. Cardiovasc Intervent Radiol. 2014 Feb;37(1):85-93. doi: 10.1007/s00270-013-0626-y. Epub 2013 May 24. PMID 23703667